CLINICAL TRIAL: NCT00794651
Title: Development of a Bedside Pain Assessment Kit for Evaluating Effectiveness of Drugs for Osteoarthritis
Brief Title: Osteoarthritis Bedside Testing Kit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Analgesic Solutions (Industry)
Responsible Party: Nathaniel Katz, MD, Analgesic Research, LLC
Other Study IDs: AR_08_MK_01
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2008-11

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; testing kit; knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OA: moderate to severe osteoarthritis of the knee

SUMMARY:
Develop and test a bedside testing kit for evaluating pain and symptoms of osteoarthritis

DETAILED DESCRIPTION:
Conduct a Focus group of subjects with painful osteoarthritis of the knee to evaluate potential kit for acceptability to subjects and investigators, and usability, clarity of instructions, appropriateness of the data capture, simplicity, subject and investigator burden, and overall impressions of the procedures.

Conduct a reliability and usability study with subjects with painful osteoarthritis of the knee to determine Intra-rater reliability, Inter-rater reliability, Kit reliability.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 50 years of age or older and has osteoarthritis of the knee.
* Subject is able to communicate meaningfully in English and comply with all study procedures.
* Subject is willing to voluntarily sign and date an informed consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to the conduct of any study-specific procedures.
* Subject has experienced a minimum duration of pain of at least 6 months.
* For each of the last 15 days, pain level has remained at least a 3 on a Pain Intensity Numerical Rating (P-NRS) scale from 0 to 10; 0 means "no pain" and 10 means "worst pain imaginable".
* Subject is ambulatory.
* Subject has a primary diagnosis of osteoarthritis of the knee by medical history.
* Subject must be willing to abstain from any pain medicine for 12 hours prior to the study.

Exclusion Criteria:

* • Subject is pregnant and/or breast-feeding.

  * Subject has a medical condition, other than OA, that is not well-controlled with treatment; or the subject has any clinically significant condition that would, in the opinion of the investigator, preclude study participation or interfere with the assessment of pain and other symptoms of OA.
  * Subject is not able to hold a stylus or pen.
  * Subject is not able to read a computer screen.
  * Subject has any chronic pain syndrome (e.g., fibromyalgia) that, in the investigator's opinion, would interfere with the assessment of pain and/or other symptoms of OA.
  * In the judgment of the investigator, the subject has a psychiatric or psychological disorder that would interfere with the completion of the study, confound the study results or pose patient risk.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: moderate to severe osteoarthritis of the knee .
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-05 (Estimated); Study Completion 2009-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Katz, MD, Principal Investigator — Analgesic Research; Thomas A Eaton, PhD, Study Director — Analgesic Research
Locations (1):
- Analgesic Research, LLC, Needham, Massachusetts, United States